CLINICAL TRIAL: NCT02206971
Title: Biomarker Feedback for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008NT001 (1203M11223)
Record Dates: First submitted 2014-07-30; First posted 2014-08-01 (Estimated); Last update posted 2020-01-10 (Actual); Status verified 2020-01

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback Group (Active Comparator): receive a Smoking Cessation Manual, the opportunity for smoking cessation counseling on the phone, and urine analyses feedback via the mail plus a phone call to discuss the information
  Interventions: Other: urine analyses feedback
- Standard Care (No Intervention): receive a Smoking Cessation Manual and the opportunity for smoking cessation counseling on the phone

INTERVENTIONS:
Other: urine analyses feedback — biomarker feedback report regarding the urine sample analyzed for the tobacco chemicals, cotinine, nicotine and NNAL
  Arms: Feedback Group

SUMMARY:
The purpose of this study is to examine the impact of providing light smokers with feedback about their health, including exposure to tobacco-related chemicals.

DETAILED DESCRIPTION:
The smoking pattern among adults in the US is undergoing a remarkable change. A substantial proportion of smokers are now light smokers (smoke ≤ 10 cigarettes per day), yet little is known about how to help light smokers quit. The prevalence of light smoking is high (~50%) among African Americans (AAs) who compared to other groups have high cotinine levels, are less successful quitting smoking, and experience disproportionately higher smoking-related cancers. Because light smokers often think that smoking fewer cigarettes a day is safe, a potential smoking cessation strategy is therefore to provide light smokers with feedback on biomarkers of tobacco exposure and increased cancer risk. The objective of this proposal is to develop and pilot test a biomarker risk assessment intervention to enhance smoking cessation for AA light smokers. The proposal builds on our previous work that shows that light smokers have 1) difficulty quitting smoking, 2) lower perceived health risks, but high levels of biomarkers (e.g. cotinine). This study will occur in 2 phases. Phase 1 will utilize focus groups to examine prevailing knowledge, attitudes, and beliefs about biomarkers as well as preferences about how participants would like to receive biomarker feedback (BF; e.g. by mail, phone, in-person). In Phase 2, data from the focus groups will be used to develop a (BF) intervention for light smokers. The new intervention will undergo further feasibility evaluation among 60 adult light smokers. Outcomes in Phase 2 will include process measures, (e.g. perceived usefulness, acceptance, and adherence) and changes in biomarker values with smoking reduction or cessation. By the end of the proposed pilot study, we expect to have developed a replicable, feasible, and acceptable BF intervention that will be ready for efficacy testing in a large clinical trial for smoking cessation or smoking reduction. The aims of the application are to: 1) Examine the prevailing knowledge, attitudes, beliefs, and preferences about BF for smoking cessation among AA light smokers; 2) Develop a BF intervention for smoking cessation among AA light smokers; and 3) Test the feasibility of a BF intervention for smoking cessation in AA light smokers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female cigarette smokers, 18-75 years
* Smoked an average of less than 10 cigarettes per day during past month
* A personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* Only one subject per household may participate
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
urinary cotinine level | week 0, week 8, week 26
  changes to biomarker levels with smoking reduction or cessation

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States